CLINICAL TRIAL: NCT05720338
Title: Is Intraperitoneal Drainage Necessary Following Distal Pancreatectomy: A Randomized Control Trial
Brief Title: Is Intraperitoneal Drainage Necessary Following Distal Pancreatectomy?
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6222
Record Dates: First submitted 2023-01-27; First posted 2023-02-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Cyst of Pancreas; Pancreatectomy; Pancreas Neoplasm
Keywords: Pancreatic neoplasm
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of care (Active Comparator): Intraperitoneal drain will be placed near the pancreatic resection margin, which is the routine standard of care.
  Interventions: Device: 19 French Blake Drain
- Omitting Standard of Care (No Intervention): No intraperitoneal drain will be placed in the participants, which omits the routine standard of care.

INTERVENTIONS:
Device: 19 French Blake Drain — 19 French Blake Intraperitoneal Drain will be placed near the pancreatic resection margin
  Other Names: Intraperitoneal drain
  Arms: Standard of care

SUMMARY:
The goal of this clinical trial is to analyze if intraperitoneal drainage is necessary following distal pancreatectomy. This study aims to determine whether the omission of routine intraperitoneal drainage in the setting of reinforced staple technology is non-inferior to routine intraperitoneal drainage with respect to a composite post-operative complications of Grade B or C Postoperative pancreatic fistula (POPF), readmission, or organ space surgical site infection following a distal pancreatectomy.

DETAILED DESCRIPTION:
Pancreatic resections are commonly performed across the United States, yet still represent one of the most morbid abdominal operations in the country, with postoperative mortality as high as 7.7%. Distal pancreatectomy (DP) represents one of the most common approaches to pancreatic resection and is typically used for tumors of the pancreatic body or tail. This operation is known to have a high historic morbidity, with reports of overall morbidity between 12-52%. Common complications include intraabdominal abscess and surgical site infection. Postoperative pancreatic fistula (POPF) represents the most common complication following partial pancreatic resection, with rates reported with rates as high as 30% in multiple large retrospective studies. Multiple strategies to prevent postoperative pancreatic leak following distal pancreatectomy have been studied. One of the outstanding questions that remains is regarding the need for routine intraperitoneal drainage following DP, particularly since the advent of reinforced staple technology. This study aims to determine if intraperitoneal drainage is necessary following DP. This study will compare groups using a composite endpoint of complications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing a scheduled distal pancreatectomy (with or without concurrent splenectomy)
* Age ≥18 years
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients < 18 years old
* Patients who are pregnant
* Patients with a history of previous pancreatic surgery
* Patients with a history of prior gastric resection, gastric bypass or sleeve gastrectomy
* Patients with prior cystogastrostomy procedure
* Patients who have failed prior endoscopic intervention or ultrasound due to esophageal or other gastrointestinal stricture
* Patients with Type 3 or Type 4 Paraesophageal Hernia noted either on pre-operative imaging or intra-operatively
* Patients undergoing concurrent resection of organs other than the pancreas or spleen or gallbladder
* Patients who undergo oversewing of the pancreatic transection margin
* Patients with unexpected intraoperative bleeding or adhesive disease which deem it unsafe to proceed without an intraabdominal drain
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint comparison | Within 90 days of surgery
  Comparison between groups using a composite endpoint of complications that includes presence of Grade B POPF
Composite endpoint comparison | Within 90 days of surgery
  Comparison between groups using a composite endpoint of complications that includes presence of Grade C POPF
Composite endpoint comparison | Within 90 days of surgery
  Comparison between groups using a composite endpoint of complications that includes Readmission
Composite endpoint comparison | Within 90 days of surgery
  Comparison between groups using a composite endpoint of complications that includes presence of Organ Space Surgical Site Infection

SECONDARY OUTCOMES:
Rates of endoscopic drainage vs percutaneous drainage of Grade B POPF | 90-day post operative time point
  Rates of drainage based off of the Grade B Postoperative pancreatic fistula
Quality of Life Score | At day 14 postoperative
  Post-operative Quality of Life score using the PROMIS-10 Global Health
Quality of Life Score | At day 14 postoperative
  Post-operative Quality of Life score using the PROMIS-10 Physical Function
Quality of Life Score | At day 14 postoperative
  Post-operative Quality of Life score using the original Drain Quality of Life scale
Quality of Life Score | At day 90 postoperative
  Post-operative Quality of Life score using the PROMIS-10 Global Health
Quality of Life Score | At day 90 postoperative
  Post-operative Quality of Life score using the PROMIS-10 Physical Function
Quality of Life Score | At day 90 postoperative
  Post-operative Quality of Life score using the original Drain Quality of Life scale
Hospital Length of Stay | 90-day post operative time point
  Measurement of the difference in Hospital Length-of-Stay based on intraperitoneal drainage after DP
Cost analysis for overall healthcare costs | At day 90 postoperative
  Cost analysis for overall healthcare costs associated with both methods of postoperative care

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simon, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No